CLINICAL TRIAL: NCT03862976
Title: Antepartum Cardiotocography With and Without Computer Analysis in High Risk Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 371/18
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computerized cardiotocography (Experimental): computerized cardiotocography
  Interventions: Diagnostic Test: computerized cardiotocography
- standard cardiotocography (Active Comparator): standard cardiotocography non stresstest
  Interventions: Diagnostic Test: computerized cardiotocography

INTERVENTIONS:
Diagnostic Test: computerized cardiotocography — computerized cardiotocography (C-CTG)

SUMMARY:
Electronic fetal hear rate monitoring (EFM), or cardiotocography (CTG), records changes in fetal heart rate and their temporal relationship to uterine contraction. It has been developed with the aim of detecting fetal hypoxia during labor and hence to prevent metabolic acidosis. Despite being the standard for intrapartum management, this technique, significantly increase the operative delivery rate, and is associated only with less seizures as neonatal benefit. Another concern is also the variability in the interpretation.

Several techniques have been studied in order to decrease the high false positive rate. Fetal ST waveform analysis (STAN) has been studied combined with CTG. A recent meta-analysis of randomized trials, however, showed that STAN during labor did not improve perinatal outcomes or decrease operative delivery rates, except for a 9% decrease in operative vaginal delivery.Comparisons of visual and computerized interpretation of EFM have also been reported. However, whether or fetal monitoring with computer analysis improve perinatal outcomes is still subject of debate.

Thus, we aim to evaluate whether intrapartum fetal monitoring with computer analysis increase the incidence of obstetric intervention when compared with visual analysis through a single-center randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton gestation
* 18 years to 50 years
* High risk pregnancies: DM, or GDM, or hypertension, or preeclampsia

Exclusion Criteria:

- IUGR

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 28 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
cesarean section | at the time of delivery
  incidence of cesarean section

SECONDARY OUTCOMES:
gestational age at delivery | at the time of delivery
  week of delivery
admission to neonatal intensive care unit | at the time of delivery
  admission to neonatal intensive care unit
birth weight | at the time of delivery
  neonatal birth weight at delivery
APGAR score at delivery | at the time of delivery
  APGAR score at delivery
neonatal death | 28 days of live of the neonate
  death of a live neonates within 28 days of life

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
not planned